CLINICAL TRIAL: NCT00530556
Title: Effect of Zolpidem vs Placebo on Insomnia and Daytime Function in Patients With Insomnia Associated With Osteoarthritis
Brief Title: Insomnia and Daytime Function in Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: L_8445
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: zolpidem

SUMMARY:
To assess the efficacy and safety of zolpidem at doses up to 10 mg compared to placebo in patients with insomnia associated with osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Patients that are male or female aged 45 years or older.
* Patients having given their written informed consent prior to participating in the trial.
* Patients who have had OA of the knee or hip for at least 6 months, as diagnosed using the American College of Rheumatology Classification Criteria for Osteoarthritis.
* Patients who, based on historical data, developed insomnia together with or after development of arthritic symptoms and presently have difficulty in maintaining sleep or have non-restorative sleep for at least three months preceding study entry and have difficulties with daytime activities because of problems with sleeping.
* Patients who, based on historical data, experience sleep disturbance at least 3 nights per week.
* Patients must have a score of greater than 1 on the Likert Pain Scale within two weeks of study participation while taking pain medication
* Patients must have been on a stable dosing regimen of analgesic/anti-inflammatory medication for one month prior to study entry and agree to maintain the dose throughout the study. Patient must agree not to exceed 4000 mg (i.e., 1000 mg acetaminophen, 4 times per day) as rescue medication in case of unexpected arthritis pain. Acetaminophen is the only rescue medication allowed in addition to the patient's stable dosing regimen.

Exclusion Criteria:

* Female patients that are pregnant or are breast-feeding.
* Patients with reproductive potential not implementing adequate contraceptive measures.
* Patients with mental disorders or who cannot be relied upon to understand the trial requirements and comply with the treatment regimen.
* Patients that are shift workers or have required a change in their regular sleep schedule by at least three hours within the last three months.
* Patients that have been treated for insomnia within 2 years prior to the onset of osteoarthritis.
* Patients that have a history of recurrent major depressive disorder over the last 3 years or any single episode of major depression over the last 2 years.
* Patients having a history of seizures or other significant neurological diseases.
* Patients with a history of myasthenia gravis.
* Patients that have had serious head injury within the past 10 years.
* Patients with insulin dependent diabetes poorly controlled in the opinion of the investigator.
* Patients who have had a stroke or myocardial infarction in the 6 months before the screening visit.
* Patients with unstable angina or severe heart failure.
* Patients with a history of significant impairment of any organ system that could impair the ability of the patient to participate in the study.
* Patients with abnormal clinical laboratory tests judged by the Investigator to require clinical intervention.
* Patients that fail to complete at least 3 of 7 consecutive nights and days (day must follow night to be consecutive) on their Evening and Morning Questionnaires during the screening period and have not satisfied the following:

  1. scored 2 or greater on the Evening Questionnaire, AND
  2. Slept a total of less than 6 hours, as determined by:

a Wake Time after Sleep Onset of greater than 1 hour, and/or having time to fall asleep (sleep latency) of 45 minutes or greater.

* Patients that have used any drug (e.g. beta-blockers, antihistamines) and subsequently reported significant CNS side effects.
* Patients with a history of hypersensitivity/exaggerated drug response to sedative/hypnotic drugs (allergic or paradoxical), including zolpidem.
* Patients with a history of sleep apnea or current signs/symptoms associated with sleep apnea
* Patients with a history of symptoms compatible with diagnosis of periodic leg movement or restless legs syndrome.
* Patients with a history of cancer within the last 5 years or that have suspected neoplastic disease (with the exception of nonmelanomatous skin cancer).
* Patients that are taking any drugs of abuse or psychotropic drugs (including, but not limited to antidepressants, antipsychotics, or anxiolytics) or drugs with demonstrated effects on sleep-wake function (including, but not limited to herbal supplements, diphenhydramine, and theophylline).
* Patients that have used over-the-counter sleep medication within seven days prior to study entry. Prescription sleep medications must have been discontinued at least 7-25 days prior to study entry, depending upon the half-life of the particular compound.
* Patients who have taken investigational drugs within 30 days of the screening visit.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2003-03; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Patient's Global Impression of Therapy of Insomnia

SECONDARY OUTCOMES:
Clinical Global Impression of Insomnia,Sleep-related outcome measures from Morning Questionnaire, Daytime Functioning Life Event Questionnaire Pain Impact Questionnaire Use of rescue medications

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi